CLINICAL TRIAL: NCT05464108
Title: Validation the Artificial Intelligence System for Automatic Evaluation of the Extent of
Brief Title: Validation the Artificial Intelligence System for Automatic Evaluation of the Extent of Intestinal Metaplasia
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Other Study IDs: 2022SDU-QILU-111
Record Dates: First submitted 2022-07-08; First posted 2022-07-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2023-12

CONDITIONS: Intestinal Metaplasia of Gastric Mucosa; Artificial Intelligence; Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — When a gastric mucosal lesion is found using IEE , endoscopist will take biopsy for histology examination. In addition, random biopsies to ensure at least four biopsies from the gastric antrum and body to cauculate the OLGIM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Gastric intestinal metaplasia observed by IEE: Get pictures from gastric antrum body and angle by image-enhanced endoscopy in order to calculate the EGGIM score.
  Interventions: Diagnostic Test: The diagnosis of Artificial Intelligence and endosopists

INTERVENTIONS:
Diagnostic Test: The diagnosis of Artificial Intelligence and endosopists — Endosopists and AI will assess the EGGIM score independently when the patients is eligible. In addition, they can not see the OLGIM score of the patients.

SUMMARY:
The operative link on gastric intestinal metaplasia assessment (OLGIM) staging systems using biopsy specimens were commonly used for histological assessment of gastric cancer risk. But its clinical application is limited for at least biopsy samples. The endoscopic grading system (EGGIM) has been shown a significant correlation with the OLGIM. The investigators designed a computer-aided diagnosis program using deep neural network to automatically evaluate the extent of IM and calculate the EGGIM scores in endoscopy examination. This study is aimed at exploring the relevance of the EGGIM scores automatically evaluated by Artificial Intelligence and OLGIM scores.

DETAILED DESCRIPTION:
Gastric intestinal metaplasia(GIM) is an important stage in the gastric cancer(GC). The operative link on gastric intestinal metaplasia assessment (OLGIM) staging systems using biopsy specimens were commonly used for histological assessment of gastric cancer risk. However, its need to take at least 4 biopsies is not clinically feasible. The endoscopic grading system (EGGIM) has been shown a significant correlation with the OLGIM. An EGGIM score of 5 was the best cut off value for identifying OLGIM stage III/IV patients. The investigators have designed a computer-aided diagnosis program using deep neural network to automatically evaluate the extent of IM and calculate the EGGIM scores in endoscopy examination. This study is aimed at exploring the relevance of the EGGIM scores automatically evaluated by Artificial Intelligence and OLGIM scores.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 40-75 years who undergo the IEE examination

Exclusion Criteria:

* patients with severe cardiac, cerebral, pulmonary or renal dysfunction or psychiatric
* disorders who cannot participate in gastroscopy
* patients with previous surgical procedures on the stomach
* patients with contraindications to biopsy
* patients who refuse to sign the informed consent form

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who receive the gastrointestinal endoscopy examination and screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of AI model to diagnose extensive intestinal metaplasia (OLGIM stage III/IV) by calculating the EGGIM score | 2 years
  A scale for endoscopic grading of gastric intestinal metaplasia (EGGIM) varies from 0 (normal endoscopy with no areas suggestive of intestinal metaplasia) to 10 (diffuse metaplasia in all gastric areas). Five different areas were considered (two areas in the antrum, two in the corpus, and one in the incisura). Each area was scored 0 (no intestinal metaplasia), 1 (focal intestinal metaplasia, ≤30 % of the area), or 2 points (extensive intestinal metaplasia in that area, > 30 % of the area), giving a possible total of 10 points. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients.

SECONDARY OUTCOMES:
Accuracy of experienced endoscopists to diagnose extensive intestinal metaplasia (OLGIM stage III/IV) by calculating the EGGIM score | 2 years
  A scale for endoscopic grading of gastric intestinal metaplasia (EGGIM) varies from 0 (normal endoscopy with no areas suggestive of intestinal metaplasia) to 10 (diffuse metaplasia in all gastric areas). Five different areas were considered (two areas in the antrum, two in the corpus, and one in the incisura). Each area was scored 0 (no intestinal metaplasia), 1 (focal intestinal metaplasia, ≤30 % of the area), or 2 points (extensive intestinal metaplasia in that area, > 30 % of the area), giving a possible total of 10 points. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients.
Accuracy of inexperienced endoscopists to diagnose extensive intestinal metaplasia (OLGIM stage III/IV) by calculating the EGGIM score | 2 years
  A scale for endoscopic grading of gastric intestinal metaplasia (EGGIM) varies from 0 (normal endoscopy with no areas suggestive of intestinal metaplasia) to 10 (diffuse metaplasia in all gastric areas). Five different areas were considered (two areas in the antrum, two in the corpus, and one in the incisura). Each area was scored 0 (no intestinal metaplasia), 1 (focal intestinal metaplasia, ≤30 % of the area), or 2 points (extensive intestinal metaplasia in that area, > 30 % of the area), giving a possible total of 10 points. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients.
Inter-observer agreement among experienced endoscopists in identifying the EGGIM scores | 2 years
  A scale for endoscopic grading of gastric intestinal metaplasia (EGGIM) varies from 0 (normal endoscopy with no areas suggestive of intestinal metaplasia) to 10 (diffuse metaplasia in all gastric areas). Five different areas were considered (two areas in the antrum, two in the corpus, and one in the incisura). Each area was scored 0 (no intestinal metaplasia), 1 (focal intestinal metaplasia, ≤30 % of the area), or 2 points (extensive intestinal metaplasia in that area, > 30 % of the area), giving a possible total of 10 points. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients.
Inter-observer agreement among inexperienced endoscopists in identifying the EGGIM scores | 2 years
  A scale for endoscopic grading of gastric intestinal metaplasia (EGGIM) varies from 0 (normal endoscopy with no areas suggestive of intestinal metaplasia) to 10 (diffuse metaplasia in all gastric areas). Five different areas were considered (two areas in the antrum, two in the corpus, and one in the incisura). Each area was scored 0 (no intestinal metaplasia), 1 (focal intestinal metaplasia, ≤30 % of the area), or 2 points (extensive intestinal metaplasia in that area, > 30 % of the area), giving a possible total of 10 points. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients.

CONTACTS AND LOCATIONS:
Overall Officials: yanqing Li, MD, PHD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastrology, QiLu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No